CLINICAL TRIAL: NCT03238456
Title: Weaving an Islander Network for Cancer Awareness, Research and Training (WINCART): Technology & Smoking Cessation for Late Adolescent/Young Adult Pacific Islanders
Brief Title: Smoking Cessation for Young Adult Pacific Islanders: Motivating Pacifika Against Cigarettes and Tobacco
Acronym: MPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Claremont Graduate University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: U54CA153458 (NIH); U54CA153458 (NIH)
Record Dates: First submitted 2017-07-21; First posted 2017-08-03 (Actual); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Tobacco Use; Tobacco Smoking; Tobacco Use Cessation; Smoking; Smoking Cessation; Smoking, Cigarette
Keywords: Pacific Islander; Native Hawaiian; NHPI; Tobacco Health; Tobacco Use; Tobacco Smoking; Tobacco Use Cessation; Smoking Cessation; Smoking; Cigarette Use; Young Adult
MeSH Terms: conditions — Tobacco Use; Tobacco Smoking; Tobacco Use Cessation; Smoking; Smoking Cessation; Cigarette Smoking | interventions — Tobacco Products

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention entitled Motivating Pacifika Against Cigarettes and Tobacco (MPACT) was implemented for eight weeks starting on the quit date that the participant chose with their assigned coach during the baseline assessment. At the baseline assessment, each participant watched an introductory video that described the online smoking cessation program. The online program was accessed through the participant's Facebook account. The program included eight education modules and a forum. Participants also received automated daily text messages to provide support and encouragement during the quitting process.
  Interventions: Behavioral: Motivating Pacifika Against Cigarettes and Tobacco
- Control (No Intervention): Participants in the control group set a quit date within two weeks of their baseline assessment and watched an introductory video that described the smoking cessation program. They received one text message every other week over a period of eight weeks following the quit date. The messages were delivered by a web-based system not connected to the online intervention program. Participants were also given a handout listing local tobacco cessation and education resources, a link to a generic online smoking cessation program, a fact sheet on smoking and tobacco use among PI young adults, and a quit kit containing chewing gum and a stress ball.

INTERVENTIONS:
Behavioral: Motivating Pacifika Against Cigarettes and Tobacco — Participants received one encouraging text message per day prior to their quit date. During the intervention, they received daily text messages with decreasing frequency per week. Participants were also able to craft personal text messages. On-demand text messages were optional and could be requested by texting key words to the program hotline.
  The online MPACT program allowed participants to access eight educational modules and a forum where they could communicate with other participants. The modules focused on different aspects of quitting smoking, such as how to deal with withdrawal symptoms, triggers of tobacco use, and stress. Participants were limited to one module per day in order to increase the duration of exposure to the program. Upon completion, participants no longer received text messages but they were still able to access the educational modules, forum, and on-demand text messages.
  Other Names: MPACT
  Arms: Intervention

SUMMARY:
The current study aimed to test a culturally tailored program designed to help Pacific Islanders (PIs) between the ages of 18 and 30 quit smoking cigarettes by using a randomized controlled trial design with one intervention group and one control group.

DETAILED DESCRIPTION:
This randomized control trial (RCT) consisted of a baseline assessment (Wave 0) and three follow-up assessments (Waves 1-3). Follow-up assessments were conducted at 2 months, 5 months, and 8 months after the baseline assessment. The objective of the study was to test a culturally-tailored online program designed to help PI young adults quit smoking cigarettes. The online program contained (1) personalized, automated text messages, (2) interactive, online educational modules, and (3) an online forum.

Hypotheses for this study include:

1. Participants in the intervention program tailored to PIs would have significantly higher rates of abstinence, lower rates of relapse, and lower smoking frequency and intensity at each follow-up time point than those in the standard intervention program.
2. Participants with impaired affective decision capacity (low scores on Iowa Gambling Task (IGT)) would benefit more from the tailored intervention program than participants with normal affective decision capacity (high IGT scores).
3. Effects from the tailored intervention program would be more pronounced among participants with particular dispositional phenotypes (depression, hostility, impulsivity) and baseline severity of tobacco addiction (nicotine dependence).
4. High-intensity users of the tailored intervention program would be more successful than low intensity users in reducing the frequency and intensity of cigarettes smoked.
5. The tailored intervention program would have greater success at engaging and retaining participants than the standard intervention program.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified as Native Hawaiian or Pacific Islander
* Between the ages 18 and 30
* Lived in Southern California
* Would be living in Southern California for the next year
* Owned a cell phone with a text messaging plan
* Had access to a computer with internet for at least 2 hours per week
* Smoked daily or most days of the week (>3 days)
* Smoked at least 100 cigarettes in lifetime

Exclusion Criteria:

• Was currently using another smoking cessation method

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 278 (Actual)
Dates: Start 2013-07-11 (Actual); Primary Completion 2014-12-03 (Actual); Study Completion 2015-05-31 (Actual)

PRIMARY OUTCOMES:
Number of cigarettes smoked in last 30 days | 8 months
  How many cigarettes has the participant smoked in the last 30 days?
Cigarette smoked in past 7 days | 8 months
  Has the participant smoked a cigarette in the past 7 days?
Cigarette smoked in past 24 hours | 8 months
  Has the participant smoked a cigarette in the past 24 hours?
Expired carbon monoxide (CO) | 8 months
  Biomarker validation (expired CO) of self-reported tobacco use

SECONDARY OUTCOMES:
Number of cigarettes smoked in last 30 days | 2 months
  How many cigarettes has the participant smoked in the last 30 days?
Number of cigarettes smoked in last 30 days | 5 months
  How many cigarettes has the participant smoked in the last 30 days?
Cigarette smoked in past 7 days | 2 months
  Has the participant smoked a cigarette in the past 7 days?
Cigarette smoked in past 7 days | 5 months
  Has the participant smoked a cigarette in the past 7 days?
Cigarette smoked in past 24 hours | 2 months
  Has the participant smoked a cigarette in the past 24 hours?
Cigarette smoked in past 24 hours | 5 months
  Has the participant smoked a cigarette in the past 24 hours?
Expired carbon monoxide (CO) | 2 months
  Biomarker validation (expired CO) of self-reported tobacco use
Expired carbon monoxide (CO) | 5 months
  Biomarker validation (expired CO) of self-reported tobacco use

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Claremont Graduate University, Claremont, California
  - California State University Fullerton, Fullerton, California

IPD SHARING:
Plan to Share IPD: Yes
De-identified datasets with individual participant data will be provided by the Principal Investigator upon request. All data sharing requests will be reviewed and approved by the Office of Research and Sponsored Programs at Claremont Graduate University and the WINCART2 Center Steering Committee.